CLINICAL TRIAL: NCT07052747
Title: Periodontal Health and Orthodontic Mini-screws: A Cross-sectional Study
Brief Title: Periodontal Effects of Orthodontic Mini-Screws
Status: Completed | Type: Observational
Sponsor: Dr. Mehmet Selim Yildiz (Other)
Responsible Party: Sponsor-Investigator, Dr. Mehmet Selim Yildiz, Assistant Professor, Dr., Altinbas University
Organization: Altinbas University (Other)
Other Study IDs: 2024/30
Record Dates: First submitted 2025-06-29; First posted 2025-07-07 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-06

CONDITIONS: Dental Implantation; Peri-implant Mucositis; Orthodontic Anchorage Procedures; Gingival Inflammation and Bleeding
MeSH Terms: conditions — Gingivitis; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical periodontal assessment — Comprehensive site-level and full-mouth evaluations of periodontal parameters, including plaque index (PI), gingival index (GI), probing pocket depth (PPD), recession depth (RD), bleeding on probing (BOP), keratinized tissue width (KTW), mucosal phenotype, mucosal redness (MR), mucosal discomfort (MD), and torque gauge (TG) measurements.

SUMMARY:
Orthodontic mini-screws (TADs) are commonly used to provide temporary anchorage and prevent unwanted tooth movement during orthodontic treatment. Their clinical success largely depends on their ability to remain stable under functional orthodontic loads. Stability is assessed in two phases: primary stability, which reflects immediate mechanical retention in bone, and secondary stability, which results from biological remodeling and healing over time. Multiple factors such as age, gender, bone characteristics, screw dimensions, and force magnitude may influence screw stability.

Recent studies suggest that local inflammation around mini-screws, similar to peri-implantitis in dental implants, can compromise bone integrity and lead to screw failure. Inadequate oral hygiene and the absence of keratinized tissue at the insertion site are among the key risk factors associated with inflammation and soft tissue complications. Unlike traditional implants, mini-screws are often inserted at variable intraoral locations and subject to angular force vectors, which may further impact surrounding periodontal tissues.

This cross-sectional clinical study aims to evaluate the effects of orthodontic mini-screw placement on general oral health and periodontal tissue status. The study will investigate site-specific and full-mouth periodontal parameters and explore potential associations between mini-screw stability, soft tissue characteristics, and signs of mucosal inflammation.

DETAILED DESCRIPTION:
Orthodontic mini-screws, also known as temporary anchorage devices (TADs), have become an integral component of modern orthodontic therapy, enabling controlled tooth movement without relying on patient compliance. For optimal clinical success, these devices must maintain mechanical stability throughout the treatment period. Stability is commonly categorized into two types: primary stability, which represents the initial mechanical engagement of the screw with cortical bone, and secondary stability, which depends on bone remodeling and healing processes occurring over time.

Despite their clinical utility, mini-screws are prone to several biological and mechanical challenges that may compromise their stability. Factors such as patient age, gender, cortical bone thickness, screw dimensions, insertion torque, and the magnitude and direction of orthodontic forces are known to affect outcomes. Moreover, local inflammatory responses-particularly in the presence of poor oral hygiene or non-keratinized soft tissue-can lead to tissue breakdown and mini-screw failure. These inflammatory reactions resemble peri-implantitis observed in dental implants and are thought to result in marginal bone loss, especially around the neck of the mini-screw.

Given the biomechanical complexity and variability in intraoral placement, orthodontic mini-screws may provoke localized periodontal changes, even in periodontally healthy individuals. However, limited data are available on how these devices influence surrounding periodontal tissues at both the site level and full-mouth level, particularly during the early healing phase after placement.

This cross-sectional clinical study aims to evaluate the relationship between orthodontic mini-screws and periodontal health three months after screw placement. A total of 132 systemically healthy, non-smoking patients with 160 mini-screw insertions will be included. Clinical parameters such as plaque index (PI), gingival index (GI), probing pocket depth (PPD), recession depth (RD), bleeding on probing (BOP), keratinized tissue width (KTW), supracrestal tissue height (STH), transmucosal soft tissue thickness (phenotype), mucosal redness (MR), and mucosal discomfort (MD) will be measured both site-specifically and at the full-mouth level. In addition, torque gauge (TG) measurements will be used to assess mechanical stability of the mini-screws.

The study aims to identify whether site-specific inflammation and soft tissue characteristics correlate with decreased implant stability or patient-reported discomfort. Results may provide valuable insights into the biological response of periodontal tissues to TADs and help improve clinical protocols for their placement, monitoring, and maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals; non-smokers; patients undergoing fixed orthodontic treatment requiring mini-screw anchorage; periodontally healthy (bleeding on probing <10%); no clinical signs of gingival inflammation at the time of mini-screw placement; provided written informed consent.

Exclusion Criteria:

* History of systemic disease (e.g., diabetes, immunosuppression); current use of antibiotics, corticosteroids, or other medications affecting periodontal health; history of radiation therapy in the head and neck region; poor oral hygiene or visible plaque accumulation at baseline; pregnant or breastfeeding women; presence of active periodontal disease (e.g., PPD >3 mm, BOP >10%); previous orthodontic mini-screw failure in the same site.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study included patients who had been treated with orthodontic mini implants at the Department of Orthodontics, Faculty of Dentistry, Altinbas University. A total of 132 patients were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth (PPD) | 3 months after mini-screw placement
  Mean PPD measured at six sites around each of the two teeth adjacent to the mini-screw, using a UNC-15 periodontal probe. Values are averaged per site to assess localized periodontal response. This measurement also done for full-mouth teeth.
Plaque Index (PI) | 3 months after mini-screw placement
  Plaque accumulation assessed visually on the buccal and lingual surfaces of teeth adjacent to the mini-screw and for full-mouth teeth using the Löe and Silness Index. Values averaged across sites.
Gingival Index (GI) | 3 months after mini-screw placement
  Gingival inflammation assessed using the Löe and Silness Gingival Index at the six surfaces of the adjacent teeth and full mouth seperately. Scores averaged to evaluate site-specific soft tissue response.
Bleeding on Probing (BOP) | 3 months after mini-screw placement
  Presence or absence of bleeding recorded at six sites per adjacent tooth and full mouth teeth immediately after gentle probing. The percentage of bleeding sites is calculated to assess inflammation.
Gingival Recession Depth (RD) | 3 months after mini-screw placement
  Distance from the cemento-enamel junction to the free gingival margin measured at six sites of adjacent teeth. Mean values indicate apical migration of the gingiva.
Mucosal Redness (MR) | 3 months after mini-screw placement
  Clinical assessment of redness in the mucosa surrounding the mini-screw, based on visual inspection. Recorded as present or absent.
Mucosal Discomfort (MD) | 3 months after mini-screw placement
  Self-reported discomfort or sensitivity around the mini-screw site, recorded during the clinical examination. Binary outcome (present or absent).
Keratinized Tissue Width (KTW) | 3 months after mini-screw placement
  Horizontal and vertical keratinized tissue widths measured using a periodontal probe in millimeters. Recorded to evaluate soft tissue protection at the site.
Supracrestal Tissue Height (STH) | 3 months after mini-screw placement
  Vertical height from the alveolar crest to the gingival margin measured at the mini-screw site using a periodontal probe. Indicates soft tissue volume and attachment.
Transmucosal Soft Tissue Thickness (Phenotype) | 3 months after mini-screw placement
  Measured using a periodontal probe to determine whether the phenotype is thick or thin. Helps assess how mucosal type influences peri-screw tissue response.
Torque Gauge (TG) Value | 3 months after mini-screw placement
  Stability of each mini-screw measured using a torque gauge. Values recorded in Newtons to assess biomechanical resistance of the screw at 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Selim YILDIZ, Asst. Prof., Principal Investigator — Altinbas University, Faculty of Dentistry
Locations (1):
- Altinbas University, Faculty of Dentistry, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Researchers can request access to the IPD by contacting Dr. Mehmet Selim Yildiz at "mehmet.yildiz2@altinbas.edu.tr or mehmetselimyildiz4@gmail.com"

REFERENCES:
- [Background] Yildiz MS, Ulutas PA, Ozenci I, Akcali A. Clinical and radiographic assessment of the association between orthodontic mini-screws and periodontal health. BMC Oral Health. 2024 Nov 14;24(1):1376. doi: 10.1186/s12903-024-05136-2. PMID 39543578
- [Background] Parmar R, Reddy V, Reddy SK, Reddy D. Determination of soft tissue thickness at orthodontic miniscrew placement sites using ultrasonography for customizing screw selection. Am J Orthod Dentofacial Orthop. 2016 Oct;150(4):651-658. doi: 10.1016/j.ajodo.2016.03.026. PMID 27692423
- [Background] Park HS, Jeong SH, Kwon OW. Factors affecting the clinical success of screw implants used as orthodontic anchorage. Am J Orthod Dentofacial Orthop. 2006 Jul;130(1):18-25. doi: 10.1016/j.ajodo.2004.11.032. PMID 16849067
- [Background] Zitzmann NU, Berglundh T, Ericsson I, Lindhe J. Spontaneous progression of experimentally induced periimplantitis. J Clin Periodontol. 2004 Oct;31(10):845-9. doi: 10.1111/j.1600-051X.2004.00567.x. PMID 15367187
- [Background] Algraffee H, Borumandi F, Cascarini L. Peri-implantitis. Br J Oral Maxillofac Surg. 2012 Dec;50(8):689-94. doi: 10.1016/j.bjoms.2011.11.020. Epub 2011 Dec 22. PMID 22197573
- [Background] Lee SJ, Ahn SJ, Lee JW, Kim SH, Kim TW. Survival analysis of orthodontic mini-implants. Am J Orthod Dentofacial Orthop. 2010 Feb;137(2):194-9. doi: 10.1016/j.ajodo.2008.03.031. PMID 20152674
- [Background] Ure DS, Oliver DR, Kim KB, Melo AC, Buschang PH. Stability changes of miniscrew implants over time. Angle Orthod. 2011 Nov;81(6):994-1000. doi: 10.2319/120810-711.1. Epub 2011 May 25. PMID 21612317
- [Background] Raghavendra S, Wood MC, Taylor TD. Early wound healing around endosseous implants: a review of the literature. Int J Oral Maxillofac Implants. 2005 May-Jun;20(3):425-31. PMID 15973954